CLINICAL TRIAL: NCT06709430
Title: Effect of Standardized Patient-Based Pain Management Program on Nursing Students' Pain Attitudes, Self-Efficacy, and Beliefs: A Double-Blind Randomized Controlled Trial
Brief Title: Effect of Standardized Patient-Based Pain Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Necibe Dağcan, Assistant Professor of Nursing, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KutahyaHSU-NECİBE-DAĞCAN-0003
Record Dates: First submitted 2024-11-07; First posted 2024-11-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Pain
Keywords: pain; nursing student; Standardized Patient; Pain Management Program; Pain Attitudes; Self-Efficacy; Beliefs
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Theoretical courses, standardized patient-based pain management laboratory practice, and clinical practice processes will be applied to students in the experimental group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Students will be randomly assigned (using online randomization software) to standardized patients group and control groups. Students will know that they are participating in the study and the interventions that will be applied to them, but they will be blinded as they will not know which group they are in. Due to the nature of the study, standardized patient and routine laboratory practices to be applied to the experimental and control groups will be applied by the first and second researchers. The research data will be collected by the third researcher who is blinded to the groups. In the statistical analysis of the data, the groups will be labeled as group 1 and group 2, and the fourth researcher will be blinded when evaluating the results. Thus, the 3rd and 4th researchers will be blinded to the study groups. In order to avoid bias in the evaluation of the results, the first and second researchers who are not blinded will not participate in any stage of the evaluation process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized Patient Group (Experimental): Students will be divided into standardized patient group and control groups. Theoretical courses, standardized patient-based pain management laboratory practice, and clinical practice processes will be applied to students in the experimental group.
  Interventions: Other: Standardized Patient Group
- Classical education group (Other): Theoretical courses, case-based pain management laboratory practice, and clinical practice processes will be applied to students in the control group.
  Interventions: Other: Classical education group

INTERVENTIONS:
Other: Classical education group — Students will be divided into standardized patient and Classical education group. Theoretical courses, standardized patient-based pain management laboratory practice, and clinical practice processes will be applied to students in the experimental group.
  Arms: Classical education group
Other: Standardized Patient Group — Students will be divided into standardized patient group and control groups. Theoretical courses, standardized patient-based pain management laboratory practice, and clinical practice processes will be applied to students in the
  Arms: Standardized Patient Group

SUMMARY:
When the studies were examined, no educational study was found to examine the effect of the standardized patient-based pain management program on the pain attitudes, self-efficacy and beliefs of nursing students. Therefore, in our study, investigators aimed to examine the effect of the standardized patient-based pain management program on the pain attitudes, self-efficacy and beliefs of nursing students. It is thought that our study results will provide evidence on pain management in undergraduate nursing education and clinics and contribute to the improvement of patient care outcomes. In addition, it is anticipated that the results of the current study will provide guidance to nurse educators for the development of pain management in nursing education and for further studies on the subject.

DETAILED DESCRIPTION:
Research Hypotheses Hypothesis 1: Standardized patient-based pain management program has an effect on nursing students' pain attitudes.

Hypothesis 2: Standardized patient-based pain management program has an effect on nursing students' pain assessment self-efficacy.

Hypothesis 3: Standardized patient-based pain management program has an effect on nursing students' pain beliefs.

This study is a double-blind randomized controlled study planned to examine the effect of a standardized patient-based pain management program on nursing students' pain attitudes, self-efficacy, and beliefs.

UNIVERSE-SAMPLE The study population will consist of students (n=157) who are studying in the 2nd year of the University in the 2024-2025 academic year, enrolled in the Basic Principles and Practices in Nursing course and continuing the course. Students who volunteer to participate in the study and meet the inclusion criteria will be randomized and numbered with the help of a computer after giving their written and verbal consent (www.randomization.com) and will be divided into two groups, each with 35 students. Group A will be called the intervention group, and Group B will be called the control group. The sample of the study was determined by the power analysis. In the G-Power statistical program, Type 1 error is 0.05, effect size is 0.80, and the sample size calculated for each group is 35, with a base power of 95%.

EDUCATIONAL MATERIALS AND DATA COLLECTION TOOLS USED IN THE RESEARCH

As educational materials in the study, for the intervention group; theoretical course content related to the subject, standardized patient and scenario will be used. For the control group, theoretical course content related to the subject and a case study in the laboratory will be used.

As data collection tools; Introductory Characteristics For Patients, Pain Beliefs Scale, Nursing Students' Attitudes Towards Pain Assessment Scale and Self-Efficacy Scale in Pain Management and Pain Management Performance Evaluation Form will be used.

COLLECTION OF DATA

The study consists of 3 stages as preparation, implementation and evaluation.

First Stage: In the first stage, the necessary preparations for the theoretical education of the study will be planned and theoretical education will be provided.

Theoretical Education, the education content regarding pain management will be prepared by the first and second researchers in line with the literature. The first researcher will explain the subject of pain management to all 2nd year nursing students (n=157) on the same day and time in 2 class hours via PowerPoint presentation and videos. Theoretical training will be carried out in 2 sessions. The first session will include definitions and types of pain, theories of pain, physiology and pathophysiology of pain. The second session will include factors affecting pain, physiological and psychological consequences of pain, communication with patients in pain and pain assessment, tools for pain assessment, and pharmacological and non-pharmacological nursing interventions in pain management.

Before and after the theoretical training, the data of the students will be collected with the Introductory Characteristics Form, Pain Beliefs Scale, Nursing Students' Attitudes Towards Pain Assessment Scale, Self-Efficacy Scale in Pain Management and Pain Management Performance Evaluation Form.

Second Stage: For the applications to be carried out with the standardized patient, the scenario will be prepared by the first and second researchers after the ethics committee permission and expert opinions will be obtained from 3 Nursing Educators who are experts in the field and the final version will be given. The same scenario will be used in the control group laboratory application but will be conducted as a case study. A university student who voluntarily participates in the study outside the nursing department and does not request a fee will serve as the standardized patient. The scenario is planned as the pain management of a patient who has undergone open heart surgery and has pain in the sternum region. The scenario will include information such as the age, marital status, occupation, education status, etc. of the standardized patient; previous diseases and hospitalization status, vital signs. The goal of the scenario is for students to diagnose, evaluate, plan and implement the patient's pain as a student nurse. Before the application, the standard patient will be trained on the purpose, method and scenario of the study, and it will be stated that he/she should not go beyond the written scenario and should not give any additional information unless the student asks. In order for the standardized patient to adapt to his/her role, the scenario will be played in a practical way as a pre-rehearsal, and the deficiencies and gaps in the scenario will be completed. Students who volunteer to participate in the study and meet the inclusion criteria will be randomized and numbered with the help of a computer after giving their written and verbal consent (www.randomization.com) and will be divided into experimental and control groups, with 35 students in each group. 2 days have been determined for laboratory/simulation applications, and the application days and times will be notified to the groups in advance.

Control group: Students in the control groups will have a case study with a scenario prepared by the faculty member responsible for each group during the laboratory application. The pain management skills of the students will be evaluated one by one by the faculty member with the "Pain Management Evaluation Form".

After laboratory applications, data will be collected from the experimental and control group students using the Pain Belief Scale, Nursing Students' Attitudes Towards Pain Assessment Scale, Self-Efficacy in Pain Management Scale and Pain Management Performance Evaluation Form.

Implementation of the Standardized Patient-Based Pain Management Program;

The stages of the implementation of the standardized patient-based pain management program are listed below:

1. Prebriefing stage: Before the simulation starts, the purpose and scope of the simulation will be explained to the students. Then, the standardized patient's history, vital signs, characteristics and scenario will be read to the students and the roles they will take in the scenario, how many minutes it will take to complete the scenario, and the goals they will reach during the scenario will be mentioned. The simulation environment and the equipment in the environment will be introduced to the students. At the same time, students will be given the opportunity to share their feelings about the simulation and their questions will be answered. In addition, in order to protect the security and integrity of the simulation environment, students will be asked not to share the simulation training with other friends.

Simulation phase: Each student's simulation application will last approximately 6-8 minutes and each student will perform the scenario once. The researcher will only observe and will not intervene until the student's application is completed. After all students in the group complete the simulation application, the debriefing session will begin.

Debriefing phase (Debriefing phase): The Plus Delta technique was used in the debriefing session. When this technique is used, 2 headings are created for the participants and positive activities are written in the plus column, and activities that can be done better or differently are written in the delta column. It is an easy method and can be easily performed with a single participant or many participants. The debriefing session will last approximately 30 minutes with the participation of all students (15-16) in the group. Students will be asked to self-assess by determining what went well or what could have been better during the simulation. At the end of the debriefing session, students will be given feedback on their performance regarding the application.

Third Phase: After theoretical and laboratory applications, students will be taken to clinical practice. During the 7-week clinical practice, all students in both the experimental and control groups will be placed in surgical clinics to provide care to patients with pain. Following the clinical practice, students' data will be collected using the Pain Belief Scale, Nursing Students' Attitudes Towards Pain Assessment Scale, Self-Efficacy in Pain Management Scale and Pain Management Performance Evaluation Form.

BIAS AND BLINDING

Students will be randomly assigned to the experimental and control groups (using online random distribution software). Students will be aware that they are participating in the study and will be blinded by the interventions that will be applied to them, but they will not know which group they are in. Due to the nature of the study, the standardized patient and routine laboratory practices to be applied to the experimental and control groups will be applied by the first and second researchers. The research data will be collected by the third researcher who is blinded to the groups. In the statistical analysis of the data, the groups will be labeled as group 1 and group 2 and the fourth researcher will be blinded when evaluating the results. Thus, the 3rd and 4th Researchers will be blinded to the study groups. To avoid bias in the evaluation of results, the unblinded first and second investigators will not participate in any stage of the evaluation process.

ELIGIBILITY:
Inclusion Criteria:

* To be a 2nd year student in the Department of Nursing
* To be registered in the Basic Principles and Practices in Nursing Course

Exclusion Criteria:

* Nursing students who did not volunteer to participate in the study,
* Having received training on pain before,
* Not participating in regular theoretical, laboratory and clinical internships during the academic period,
* Having worked or are working as a health worker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Pain Beliefs Scale mean score | up to 15 weeks
  Pain Beliefs Scale has a total of 12 items covering pain beliefs. The scale has 8 "Organic Beliefs" and 4 "Psychological Beliefs" sub-dimensions. The items in the scale are rated using a Likert-type scoring system ranging from 1 to 6 (1-always, 2-almost always, 3-often, 4-sometimes, 5-rarely, 6-never). The total score for each sub-dimension is calculated by summing the scores from the items in that sub-dimension and dividing them by the number of items in that sub-dimension. There is no cut-off point for scale scores; an increase in the score from a sub-score of the scale indicates that pain beliefs related to that test are high, while a decrease in the score indicates that pain beliefs related to that test are low. The highest score that can be obtained from the organic and psychological beliefs sub-dimensions is 6, and the lowest score is 1.

SECONDARY OUTCOMES:
Attitudes mean score | up to 15 weeks
  Nursing Students' Attitudes Towards Pain Assessment Scale: The minimum score obtained from the scale is "15" and the maximum score is "75". As the score obtained from the scale increases, the positive attitudes of nursing students towards pain assessment also increase.
Self-Efficacy mean score | up to 15 weeks
  Self-Efficacy Scale in Pain Management: The general scale score varies between min: 0 and max: 105. There is no cut-off point in the scale. It is stated that as the score increases, compliance increases.

CONTACTS AND LOCATIONS:
Overall Officials: Şenay TAKMAK, PhD, Study Director — Kütahya Health Sciences University, Faculty of Health Sciences; Burcu NAL, PhD, Study Director — Kütahya Health Sciences University, Faculty of Health Sciences; Ferzan KALAYCI EMEK, PhD (c), Study Director — Kütahya Health Sciences University, Faculty of Health Sciences
Locations (1):
- Necibe, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No